CLINICAL TRIAL: NCT06599359
Title: Intention to Leave, Job Stress, Burnout, and Job Satisfaction Among Pharmacists in Lebanon
Acronym: BLISS
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Associate Clinical and Epidemiological Professor, Lebanese University
Other Study IDs: 19/24/D
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Job Satisfaction; Burnout; Intention to Leave
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pharmacists: Employed Lebanese Pharmacists/Pharmacy Students
  Interventions: Behavioral: BLISS Questionnaire

INTERVENTIONS:
Behavioral: BLISS Questionnaire — After extensive literature review and review from the IRB of the Lebanese University. A questionnaire was developed to assess the Intention to leave, job stress, burnout, and job satisfaction among pharmacists in Lebanon
  The following sections will be considered:
  * Socio-economic characteristics
  * Work-related characteristics
  * Job stress assessment (Likert scale)
  * Burnout assessment (Likert scale)
  * Intention to Leave assessment (Likert scale)

SUMMARY:
In Lebanon, the situation of pharmacists is complicated by external factors such as economic instability and healthcare system challenges. The economic crisis has led to financial strain for many pharmacists, affecting their income and job security. Additionally, shortages of medications and medical supplies, along with high patient loads, contribute to increased job stress and burnout. Political instability adds another layer of uncertainty and stress, impacting the overall mental well-being of healthcare professionals. Recent studies emphasize the need for interventions to mitigate job stress and burnout among pharmacists. No study has comprehensively assessed these themes among pharmacists in Lebanon, especially after the COVID-19 pandemic and the consequences of the economic crisis. This study aims to test the dynamics of intention to leave, job stress, burnout, and job satisfaction among pharmacists due to their significant impact on healthcare delivery.

DETAILED DESCRIPTION:
The study aims to explore the dynamics between job stress, burnout, job satisfaction, and the intention to leave the profession among pharmacists in Lebanon. Here's a detailed description:

1. Study Overview and Purpose The research seeks to understand the complex relationships between job stress, burnout, job satisfaction, and pharmacists intentions to leave their jobs. These factors are highly significant as they directly impact the healthcare system's stability and the quality of care provided .

   Pharmacists, like other healthcare workers, face intense stress due to high workloads, long hours, and the essential nature of their responsibilities. In Lebanon, these stressors are compounded by the ongoing economic crisis, political instability, and shortages of medical supplies .
2. State of the Problem Burnout: This is characterized by emotional exhaustion, depersonalization, and a decreased sense of personal accomplishment. Burnout not only harms the mental and physical well-being of pharmacists but also leads to reduced job performance and increased errors .

   Job Satisfaction: Job satisfaction is influenced by working conditions, recognition, opportunities for growth, and interpersonal relationships. High job satisfaction is linked to better performance and lower turnover, while low satisfaction increases the likelihood of pharmacists leaving their jobs .

   External Factors: In Lebanon, pharmacists face additional pressures due to economic challenges, such as reduced income and job security, along with medication shortages and political instability . These factors worsen job stress and contribute to burnout, affecting overall job satisfaction and pushing pharmacists toward leaving the profession.
3. Research Format and Methodology (PECO) Population: Employed pharmacists and pharmacy students in Lebanon. Exposure: The changing work environment, especially after the COVID-19 pandemic and the ongoing economic crisis .

   Comparison: A questionnaire will assess the intention to leave, job stress, burnout, and job satisfaction .

   Outcomes: The study will examine correlations between the scores on job stress, burnout, and satisfaction scales and the participants' demographic characteristics
4. Questionnaire Structure Socio-economic and Work-Related Characteristics: This section gathers information about the participants' demographic and work environment details.

   Job Stress Assessment: A Likert scale is used to measure the participants' levels of job stress .

   Burnout Assessment: A Likert scale measures burnout symptoms like emotional exhaustion and depersonalization.

   Intention to Leave Assessment: This scale assesses how likely pharmacists are to leave their jobs due to stress, burnout, or dissatisfaction .
5. Study Timeline and Expected Outcomes The study began on July 15th, 2024, and data collection is ongoing. The outcomes will include a thesis, a scientific publication in a peer-reviewed journal, and potentially a presentation at an international conference .

The study will provide valuable insights into the mental health and job satisfaction of pharmacists in Lebanon, highlighting the need for interventions to reduce job stress and burnout in this critical sector.

ELIGIBILITY:
Inclusion Criteria:

* Employed Lebanese Pharmacists/Pharmacy Students
* Above 18 years
* Those agreeing to participate in the study

Exclusion Criteria:

* Unemployed pharmacists for more than one month
* Non-Lebanese
* Those with mental conditions who cannot answer the survey
* Those who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pharmacists and pharmacy students in Lebanon
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pharmacists perception | through study completion, an average of 3 months
  Correlation between the score of the intention to leave, burnout and satisfaction schemes with the participants general characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Hatem, PhD, Principal Investigator — Clinical and Epidemiological Research Laboratory, Faculty of Pharmacy, Lebanese University
Locations (2):
- Lebanon (2):
  - Pharmacy Du Liban, Beirut
  - Lebanese University, Beirut

IPD SHARING:
Plan to Share IPD: Undecided